CLINICAL TRIAL: NCT00092495
Title: A Study to Demonstrate Immunogenicity and Tolerability of Gardasil (V501) Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in Preadolescents, and To Determine End-Expiry Specifications for the Vaccine
Brief Title: Study of an Investigational Vaccine in Pre-Adolescents and Adolescents (Gardasil)(V501-016)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-016; 2004_083
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Results first posted 2010-03-08 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Cancer; Genital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Vaccines, Synthetic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): 100% Formulation qHPV Vaccine
  Interventions: Biological: V501, Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine
- 2 (Experimental): 60% Formulation qHPV Vaccine
  Interventions: Biological: V501, Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine
- 3 (Experimental): 40% Formulation qHPV Vaccine
  Interventions: Biological: V501, Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine
- 4 (Experimental): 20% Formulation qHPV Vaccine
  Interventions: Biological: V501, Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine

INTERVENTIONS:
Biological: V501, Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine — qHPV Vaccine (20, 40, 60 or 100% dose formulation) 0.5 mL intramuscular injection given at Day 1, Month 2 and Month 6.
  Other Names: V501; Gardasil

SUMMARY:
The primary purpose of the study is to determine if an investigational vaccine Gardasil (V501) with 4 components will provide an immune response and will be well tolerated in pre-adolescents and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents and pre-adolescents with no prior sexual history
* Healthy women who have an intact uterus with lifetime history of 0-4 sexual partners

Exclusion Criteria:

* Prior Human Papillomavirus (HPV) vaccination
* Prior abnormal Paps
* Prior history of genital warts

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3055 (Actual)
Dates: Start 2002-12; Primary Completion 2004-09 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Block SL, Nolan T, Sattler C, Barr E, Giacoletti KE, Marchant CD, Castellsague X, Rusche SA, Lukac S, Bryan JT, Cavanaugh PF Jr, Reisinger KS; Protocol 016 Study Group. Comparison of the immunogenicity and reactogenicity of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in male and female adolescents and young adult women. Pediatrics. 2006 Nov;118(5):2135-45. doi: 10.1542/peds.2006-0461. PMID 17079588
- [Background] Barr E, Gause CK, Bautista OM, Railkar RA, Lupinacci LC, Insinga RP, Sings HL, Haupt RM. Impact of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like particle vaccine in a sexually active population of North American women. Am J Obstet Gynecol. 2008 Mar;198(3):261.e1-11. doi: 10.1016/j.ajog.2007.09.001. PMID 18313445
- [Background] Perez G, Lazcano-Ponce E, Hernandez-Avila M, Garcia PJ, Munoz N, Villa LL, Bryan J, Taddeo FJ, Lu S, Esser MT, Vuocolo S, Sattler C, Barr E. Safety, immunogenicity, and efficacy of quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like-particle vaccine in Latin American women. Int J Cancer. 2008 Mar 15;122(6):1311-8. doi: 10.1002/ijc.23260. PMID 18000825
- [Background] Giuliano AR, Lazcano-Ponce E, Villa L, Nolan T, Marchant C, Radley D, Golm G, McCarroll K, Yu J, Esser MT, Vuocolo SC, Barr E. Impact of baseline covariates on the immunogenicity of a quadrivalent (types 6, 11, 16, and 18) human papillomavirus virus-like-particle vaccine. J Infect Dis. 2007 Oct 15;196(8):1153-62. doi: 10.1086/521679. Epub 2007 Sep 17. PMID 17955433
- [Derived] Garland SM, Ault KA, Gall SA, Paavonen J, Sings HL, Ciprero KL, Saah A, Marino D, Ryan D, Radley D, Zhou H, Haupt RM, Garner EIO; Quadrivalent Human Papillomavirus Vaccine Phase III Investigators. Pregnancy and infant outcomes in the clinical trials of a human papillomavirus type 6/11/16/18 vaccine: a combined analysis of five randomized controlled trials. Obstet Gynecol. 2009 Dec;114(6):1179-1188. doi: 10.1097/AOG.0b013e3181c2ca21. PMID 19935017
- [Derived] Majewski S, Bosch FX, Dillner J, Iversen OE, Kjaer SK, Munoz N, Olsson SE, Paavonen J, Sigurdsson K, Bryan J, Esser MT, Giacoletti K, James M, Taddeo F, Vuocolo S, Barr E. The impact of a quadrivalent human papillomavirus (types 6, 11, 16, 18) virus-like particle vaccine in European women aged 16 to 24. J Eur Acad Dermatol Venereol. 2009 Oct;23(10):1147-55. doi: 10.1111/j.1468-3083.2009.03266.x. Epub 2009 Apr 23. PMID 19453788

RESULTS

PARTICIPANT FLOW:
Groups:
- 20% Formulation qHPV Vaccine: Subjects in this group received a 20% dose formulation of the quadrivalent human papillomavirus (qHPV) vaccine at Day 1, Month 2, and Month 6.
- 40% Formulation qHPV Vaccine: Subjects in this group received a 40% dose formulation of the qHPV vaccine at Day 1, Month 2, and Month 6.
- 60% Formulation qHPV Vaccine: Subjects in this group received a 60% dose formulation of the qHPV vaccine at Day 1, Month 2, and Month 6
- 100% Formulation qHPV Vaccine: Subjects in this group received a 100% dose formulation of the qHPV vaccine at Day 1, Month 2, and Month 6.
- Extension Study: Extension Study: This group includes 12 subjects who participated in the base study and received either a partial dose formulation of the quadrivalent HPV vaccine in the base study and did not meet the protocol specified criteria for seroconversion, or subjects who, due to pregnancy, received 1 or 2 doses of the quadrivalent HPV vaccine in the base study and remained in the study through Month 7. The Extension Period began after all patients had completed the Month 7 follow-up period. Subjects designated as "Completed Period" are those who at the end of the study had received three injections of quadrivalent HPV vaccine and completed all follow-up visits. Subjects designated as "Not Completed" are those who: a) Received all three vaccinations, but did not complete follow-up; b) Did not receive all vaccinations, but completed follow-up, or c) Did not receive all vaccinations, and did not complete follow-up.
Period: Base Study Vaccination Period
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine | Extension Study
Started | 504 | 514 | 508 | 1529 | 0
With Long-term Follow-up * | 2 (Subjects received fewer than 3 doses of vaccinations and entered the long-term follow-up period) | 2 (Subjects received fewer than 3 doses of vaccinations and entered the long-term follow-up period) | 6 (Subjects received fewer than 3 doses of vaccinations and entered the long-term follow-up period) | 10 (Subjects received fewer than 3 doses of vaccinations and entered the long-term follow-up period) | 0
Without Long-term Follow-up | 34 (Subjects discontinued on or before Month 7 and did not enter the long-term follow-up period) | 20 (Subjects discontinued on or before Month 7 and did not enter the long-term follow-up period) | 28 (Subjects discontinued on or before Month 7 and did not enter the long-term follow-up period) | 73 (Subjects discontinued on or before Month 7 and did not enter the long-term follow-up period) | 0
Completed | 467 (Completed 3 vaccinations; entered the long-term follow-up or completed the study per-protocol) | 492 (Completed 3 vaccinations; entered the long-term follow-up or completed the study per-protocol) | 474 (Completed 3 vaccinations; entered the long-term follow-up or completed the study per-protocol) | 1441 (Completed 3 vaccinations; entered the long-term follow-up or completed the study per-protocol) | 0
Not Completed | 37 | 22 | 34 | 88 | 0
Not completed — Randomized Not Vaccinated | 1 | 1 | 0 | 4 | 0
Not completed — Extended | 0 | 0 | 0 | 1 | 0
Not completed — *Clinical AE | 1 | 0 | 1 | 2 | 0
Not completed — *Other reasons | 1 | 0 | 0 | 1 | 0
Not completed — *Pregnancy | 0 | 2 | 5 | 7 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 16 | 6 | 11 | 36 | 0
Not completed — Moved | 3 | 1 | 2 | 2 | 0
Not completed — Other | 1 | 1 | 0 | 2 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0 | 0
Not completed — Parent Withdrew Consent | 1 | 1 | 1 | 5 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 10 | 14 | 25 | 0
Period: Base Study Follow-up Period
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine | Extension Study
Started | 115 (Protocol amended to extend follow-up for 10-15 year old subjects to Month 12 (6 months Postdose 3)) | 125 (Protocol amended to extend follow-up for 10-15 year old subjects to Month 12 (6 months Postdose 3)) | 130 (Protocol amended to extend follow-up for 10-15 year old subjects to Month 12 (6 months Postdose 3)) | 460 (Protocol amended to extend follow-up for 10-15 year old subjects to Month 12 (6 months Postdose 3)) | 0
Completed | 112 | 122 | 126 | 446 | 0
Not Completed | 3 | 3 | 4 | 14 | 0
Not completed — Extended | 0 | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 3 | 3 | 12 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Period: Extension Study
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine | Extension Study
Started | 0 | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 0 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine | Total
Number analyzed (Participants) | 504 | 514 | 508 | 1529 | 3055
Age, Continuous [Mean (Full Range); unit: years] | 16.2 [10 to 23] | 16.5 [10 to 24] | 16.2 [10 to 23] | 15.1 [10 to 23] | 15.7 (10) [10 to 24]
Age, Customized [Number; unit: participants]
  10 to 11 Years of Age | 75 | 77 | 74 | 302 | 528
  12 to 13 Years of Age | 110 | 95 | 101 | 370 | 676
  14 to 15 Years of Age | 67 | 83 | 77 | 344 | 571
  16 to 17 Years of Age | 40 | 24 | 35 | 77 | 176
  18 to 19 Years of Age | 58 | 62 | 71 | 125 | 316
  20 to 21 Years of Age | 90 | 86 | 93 | 165 | 434
  22 to 23 Years of Age | 64 | 86 | 57 | 146 | 353
  Over 23 Years of Age | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 504 | 514 | 508 | 1019 | 2545
  Male | 0 | 0 | 0 | 510 | 510

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Seroconverted for HPV 6 by Week 4 Postdose 3
Description: Seroconversion is defined as going from seronegative to seropositive.
  Seropositivity is defined as an anti-HPV 6 titer ≥ 20 milliMerck units per milliliter (mMU/mL).
Time Frame: Week 4 Postdose 3 (Month 7)
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data. Restricted to subjects receiving 100% dosage.
Measure: Number; unit: Subjects
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 423 | 428 | 320
Subjects
  HPV 6 ≥ 20 mMU/mL | 423 | 428 | 320
  HPV 6 < 20 mMU/mL | 0 | 0 | 0
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (girls - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (boys - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

2. Primary Outcome: Geometric Mean Titer (GMT) for HPV 6 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: : Per-protocol population: subjects must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data. Restricted to subjects receiving 100% dosage.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 423 | 428 | 320
mMU/mL | 987.3 [905.0 to 1077.0] | 1116.1 [1022.7 to 1218.1] | 603.0 [548.5 to 662.9]
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (girls/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (boys/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

3. Primary Outcome: Number of Subjects Who Seroconverted for HPV 6 by Week 4 Postdose 3
Description: as for outcome 1
Time Frame: Week 4 Postdose 3 (Month 7)
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data. Restricted to female subjects 10-15 years and 16-23 years.
Measure: Number; unit: Subjects
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 372 | 391 | 364 | 743
Subjects
  HPV 6 ≥ 20 mMU/mL | 372 | 391 | 363 | 743
  HPV 6 < 20 mMU/mL | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

4. Primary Outcome: Geometric Mean Titer (GMT) for HPV 6 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 372 | 391 | 364 | 743
mMU/mL | 584.2 [526.7 to 647.9] | 704.5 [636.6 to 779.7] | 707.5 [632.5 to 791.2] | 798.4 [747.1 to 853.2]
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

5. Primary Outcome: Number of Subjects Who Seroconverted for HPV 11 by Week 4 Postdose 3
Description: Seroconversion is defined as going from seronegative to seropositive.
  Seropositivity is defined as an anti-HPV 11 titer ≥ 16 milliMerck units per milliliter (mMU/mL).
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 423 | 428 | 320
Subjects
  HPV 11 ≥ 16 mMU/mL | 423 | 428 | 320
  HPV 11 < 16 mMU/mL | 0 | 0 | 0
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (girls - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (boys - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

6. Primary Outcome: Geometric Mean Titer (GMT) for HPV 11 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 423 | 428 | 320
mMU/mL | 1264.0 [1153.2 to 1385.4] | 1396.5 [1271.4 to 1534.0] | 739.2 [665.6 to 821.0]
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (girls/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (boys/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

7. Primary Outcome: Number of Subjects Who Seroconverted for HPV 11 by Week 4 Postdose 3
Description: as for outcome 5
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 373 | 391 | 365 | 743
Subjects
  HPV 11 ≥ 16 mMU/mL | 373 | 391 | 364 | 743
  HPV 11 < 16 mMU/mL | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

8. Primary Outcome: Geometric Mean Titer (GMT) for HPV 11 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: : Per-protocol population: subjects must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data. Restricted to female subjects 10-15 years and 16-23 years.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 373 | 391 | 365 | 743
mMU/mL | 632.1 [565.2 to 706.8] | 804.7 [723.9 to 894.4] | 836.2 [743.7 to 940.2] | 1003.2 [934.0 to 1077.6]
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

9. Primary Outcome: Number of Subjects Who Seroconverted for HPV 16 by Week 4 Postdose 3
Description: Seropositivity is defined as an anti-HPV 16 titer ≥ 20 milliMerck units per milliliter (mMU/mL). Seroconversion is defined as going from seronegative to seropositive.
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number; unit: mMU/mL
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 424 | 427 | 306
mMU/mL
  HPV 16 ≥ 20 mMU/mL | 424 | 427 | 306
  HPV 16 < 20 mMU/mL | 0 | 0 | 0
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (girls - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (boys - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

10. Primary Outcome: Geometric Mean Titer (GMT) for HPV 16 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 424 | 427 | 306
mMU/mL | 4848.8 [4350.2 to 5404.5] | 5923.0 [5325.2 to 6587.9] | 2753.0 [2400.5 to 3157.3]
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (girls/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (boys/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

11. Primary Outcome: Number of Subjects Who Seroconverted for HPV 16 by Week 4 Postdose 3
Description: Seroconversion is defined as going from seronegative to seropositive.
  Seropositivity is defined as an anti-HPV 16 titer ≥ 20 milliMerck units per milliliter (mMU/mL).
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 365 | 375 | 365 | 730
Subjects
  HPV 16 ≥ 20 mMU/mL | 365 | 375 | 364 | 730
  HPV 16 < 20 mMU/mL | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.01, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

12. Primary Outcome: Geometric Mean Titer (GMT) for HPV 16 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 365 | 375 | 365 | 730
mMU/mL | 2401.1 [2084.0 to 2766.6] | 2963.3 [2593.3 to 3386.0] | 3105.3 [2692.8 to 3581.1] | 3824.6 [3504.4 to 4174.2]
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

13. Primary Outcome: Number of Subjects Who Seroconverted for HPV 18 by Week 4 Postdose 3
Description: Seroconversion is defined as going from seronegative to seropositive.
  Seropositivity is defined as an anti-HPV 18 titer ≥ 24 milliMerck units per milliliter (mMU/mL).
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 426 | 429 | 340
Subjects
  HPV 18 ≥ 24 mMU/mL | 426 | 428 | 337
  HPV 18 < 24 mMU/mL | 0 | 1 | 3
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (girls - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (boys - women) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

14. Primary Outcome: Geometric Mean Titer (GMT) for HPV 18 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: subjects must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data. Restricted to subjects receiving 100% dosage.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 10-15 Years | Boys 10-15 Years | Women 16-23 Years
Number analyzed (Participants) | 426 | 429 | 340
mMU/mL | 953.6 [857.3 to 1060.7] | 1232.9 [1105.6 to 1375.0] | 470.5 [418.5 to 528.9]
Statistical Analysis 1: Comparison: Girls 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (girls/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: Boys 10-15 Years vs Women 16-23 Years; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (boys/women) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

15. Primary Outcome: Number of Subjects Who Seroconverted for HPV 18 by Week 4 Postdose 3
Description: as for outcome 13
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 382 | 406 | 379 | 766
Subjects
  HPV 18 ≥ 24 mMU/mL | 381 | 403 | 375 | 763
  HPV 18 < 24 mMU/mL | 1 | 3 | 4 | 3
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (partial dose - full dose) must be greater than -5%; p < 0.001, Miettinen and Nurminen; Miettinen and Nurminen method for difference in proportions Miettinen and Nurminen, Stat Med 1985;4:213-26

16. Primary Outcome: Geometric Mean Titer (GMT) for HPV 18 by Week 4 Postdose 3
Time Frame: Week 4 Postdose 3 (Month 7)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | 20% Formulation qHPV Vaccine | 40% Formulation qHPV Vaccine | 60% Formulation qHPV Vaccine | 100% Formulation qHPV Vaccine
Number analyzed (Participants) | 382 | 406 | 379 | 766
mMU/mL | 544.0 [480.9 to 615.3] | 640.4 [570.5 to 718.9] | 647.5 [571.6 to 733.5] | 696.9 [641.7 to 756.8]
Statistical Analysis 1: Comparison: 20% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 2: Comparison: 40% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group
Statistical Analysis 3: Comparison: 60% Formulation qHPV Vaccine vs 100% Formulation qHPV Vaccine; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (partial dose/full dose) must be greater than 0.5; p < 0.001, ANOVA; ANOVA on natural log titer with fixed effects for region and comparison group

ADVERSE EVENTS:
Description: Adverse events were collected from subjects with follow-up.
Groups:
- 20% Formulation: Subjects in this group received a 20% dose formulation of the quadrivalent human papillomavirus (qHPV) vaccine at Day 1, Month 2, and Month 6.
- 40% Formulation: Subjects in this group received a 40% dose formulation of the quadrivalent human papillomavirus (qHPV) vaccine at Day 1, Month 2, and Month 6.
- 60% Formulation: Subjects in this group received a 60% dose formulation of the quadrivalent human papillomavirus (qHPV) vaccine at Day 1, Month 2, and Month 6.
- 100% Formulation: Subjects in this group received a 100% dose formulation of the quadrivalent human papillomavirus (qHPV) vaccine at Day 1, Month 2, and Month 6.
Arm/Group | 20% Formulation | 40% Formulation | 60% Formulation | 100% Formulation
Serious Adverse Events (participants affected / at risk) | 5/496 | 2/509 | 1/500 | 4/1498
Other Adverse Events (participants affected / at risk) | 434/496 | 426/509 | 431/500 | 1276/1498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20% Formulation (N=496) | 40% Formulation (N=509) | 60% Formulation (N=500) | 100% Formulation (N=1498)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia foetal (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20% Formulation (N=496) | 40% Formulation (N=509) | 60% Formulation (N=500) | 100% Formulation (N=1498)
Nausea (Gastrointestinal disorders) | 35 (40) | 31 (36) | 29 (35) | 65 (67)
Injection site erythema (General disorders) | 114 (157) | 116 (163) | 113 (157) | 324 (436)
Injection site pain (General disorders) | 402 (863) | 395 (881) | 395 (879) | 1184 (2535)
Injection site swelling (General disorders) | 119 (179) | 130 (201) | 121 (172) | 359 (500)
Pyrexia (General disorders) | 72 (89) | 69 (93) | 51 (59) | 196 (238)
Nasopharyngitis (Infections and infestations) | 23 (23) | 30 (36) | 30 (32) | 70 (70)
Dizziness (Nervous system disorders) | 25 (28) | 9 (13) | 19 (19) | 39 (43)
Headache (Nervous system disorders) | 127 (202) | 120 (176) | 143 (221) | 348 (490)

LIMITATIONS AND CAVEATS:
Of note, the number of subjects who completed the Vaccination Period (N=1441) is slightly higher than that specified in the publication by Block, et al (2006; N=1430). The data provided here is based on final data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.